CLINICAL TRIAL: NCT05979805
Title: Effectiveness of Motivational Interviewing and Conventional Oral Health Education (OHEc) Versus OHEc in the Prevention and Control of Dental Caries and Gingivitis in Subjects With Fixed Orthodontic Appliances. A Randomized Controlled Trial
Brief Title: Effectiveness of Two Health Education Interventions in the Prevention of Caries and Gingivitis in Orthodontic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Responsible Party: Principal Investigator, Adriana del Pilar Forero, Associate professor, Department of Oral health, Orthodontic Sciences , National University of Colombia, Universidad Nacional de Colombia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ECA 103-23
Record Dates: First submitted 2023-07-12; First posted 2023-08-07 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Dental Caries; Tooth Demineralization; Gingivitis
Keywords: Adolescent,Teenagers,Young Adult,Adult; "Motivational Interviewing"[Mesh]; "Health Education, Dental"[Mesh]; "Orthodontic Appliances"[Mesh]; "Orthodontic Appliances, Fixed"[Mesh]
MeSH Terms: conditions — Dental Caries; Tooth Demineralization; Gingivitis

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical trial open to subjects and single-blinded (investigators) of parallel groups is proposed for the evaluation of the effect of conventional educational interventions and motivational interviewing in comparison with conventional educational interventions, in the prevention of dental caries lesions and gingivitis in 94 patients aged 13 to 28 years old, who will begin corrective orthodontic treatment with fixed appliances in the postgraduate clinics of Orthodontics and Maxillary Orthopedics of the National University of Colombia.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The randomization tool of the RedCap (Research Electronic Data Capture) platform will be used. The randomizing will be performed by an independent investigator who has no contact or access to the information of the subjects, ensuring that the allocation will be blinded for the rest of the investigators. The patient will know the assigned group when he or she is scheduled to the motivational intervention, thus the study will be open to the subjects.
  The investigator who performs motivational and usual intervention is not blinded because once the patient is summoned for the application of motivational intervention, he/she will know the assigned group. Investigators who perform clinical measurements and indexes will remain blinded throughout the study by means of restricted access to the randomization instrument and general data recording of the study. The statistical data evaluator will be unaware of the allocation of the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Oral health Education (Active Comparator): Conventional oral health education and nutritional guidelines prior to the placement of fixed appliances, by means of a 5-8 minute video and instructive brochure.
  Interventions: Other: Conventional Educational interventions
- Motivational interviewing + Conventional Oral health Education (Experimental): Include the conventional oral health education of the control group and a 30 minute motivational interviewing (MI)
  Interventions: Other: Conventional Educational interventions; Behavioral: Motivational intervention

INTERVENTIONS:
Other: Conventional Educational interventions — Conventional educational methods can be verbal, written or visual and can be combined for greater understanding and effectiveness in oral health and dietary routines. The education are imparted in the first appointment of the appliances cementation by a video and oral health instruction booklet and each patient receive an oral hygiene kit. This education is repeated in month 1 and 3 after appliances cementation.
Behavioral: Motivational intervention — In addition to the conventional educational method, a motivational interviewing (MI) by Miller and Rollnick of 30 minutes will be used, with an initial script according to the stage of change in each patient in T0. The reinforcements of motivational interviewing are in month one and three after the installation of the braces, they will have the same methodology but will be focused on the aspects that in the previous session or in the clinical assessment were detected as the most important deficiencies or risk factors for the patient.
  Arms: Motivational interviewing + Conventional Oral health Education

SUMMARY:
Dental caries and gingivitis are classified by the World Health Organization (WHO) as an important public health problem due to their high prevalence and incidence worldwide despite the development of public policies to combat them. They are chronic diseases that have a severe impact in terms of pain and suffering, impairment of function and effect on quality of life. During orthodontic treatments, the most common adverse event is the appearance of dental caries lesions and gingivitis due to increased retention and change of dental biofilm composition or difficulty of removal with conventional oral hygiene techniques. Efforts to implement various conventional preventive interventions of self-care and education have not decreased their incidence, so it is necessary to implement motivational interventions to help adolescents and young adults to make positive changes in their oral health habits, which are constant and lasting and prevent and control gingivitis and caries.

DETAILED DESCRIPTION:
Dental caries and gingivitis are multifactorial diseases, however the only necessary factor, although insufficient for their development, is bacterial biofilm; brackets significantly increase its retention and limit self- cleaning mechanisms, representing a challenge in clinical practice. Motivational interventions in oral health could be an alternative to generate behavioral changes in oral health and daily self-care routines that are more sustainable over time compared to conventional education models in patients with fixed orthodontic appliances. A randomized controlled clinical trial open to subjects and single-blinded (investigators) of parallel groups is proposed for the evaluation of the effect of motivational interviewing combined with conventional oral health education (OHEc) versus OHEc, in the prevention of dental caries lesions and gingivitis. A sample size of 94 patients in total is proposed, distributed 47 in each arm of the study, with a follow-up of the cohort for six months. The baseline risk will be established before the placement of fixed appliances (T0), and a follow-up will be carried out during six months, with assessments in one (T1), three(T2) and six months (T3) after cementation, where the presence of gingivitis, caries and changes in risk variables, adverse events and adherence to conventional and motivational interventions, will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the different orthodontic postgraduate clinics of the National University of Colombia who requires treatment with fixed orthodontic appliances
* 13 years old up to 28 years of age.
* Willingness to participate in the study and signature of the informed consent form.

Exclusion Criteria:

* Patients with untreated caries lesions
* Patients with periodontal diseases or experience
* Previous orthodontics treatments
* Severe fluorosis or enamel abnormalities.
* Medical compromise or treatments generating hyposalivation or gingival enlargement
* Craniomaxillary anomalies
* Cognitive or motor disability
* Pregnancy.
* Dependence to alcohol, nicotine or psychoactive substances

Ages: 13 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Changes in ICDAS score of the caries | 6 months
  Change in incidence of caries on the vestibular and proximal surfaces by ICDAS and radiographic ICDAS in T0 (baseline),T1 (1 month),T2 (3 months) and T3 (6 months) will be censured when the patient presents the outcome, the study period ends (six months) or when the follow-up period finishes for a reason other than the event of interest being studied.
Evaluation of gingivitis | 6 months
  Changes in modification of the Silness and Löe gingival index described by Williams at T0 (baseline), T1 (one month), T2 (three months) and T3 (six months) after the start of orthodontic treatment with fixed appliances.

SECONDARY OUTCOMES:
Change of Plaque index | 6 months
  Changes in modification of the Silness and Löe index described by Williams at T0 (baseline), T1 (one month), T2 (three months) and T3 (six months) after the start of orthodontic treatment with fixed appliances.

OTHER OUTCOMES:
Adverse events | 6 months
  Measurement of possible adverse events during educational interventional at T0 (baseline), T1 (one month), T2 (three months) and T3 (six months) after the start of orthodontic treatment with fixed appliances.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Forero Niño, DDs, Principal Investigator — 111211
Locations (1):
- Universidad Nacional de Colombia, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sundararaj D, Venkatachalapathy S, Tandon A, Pereira A. Critical evaluation of incidence and prevalence of white spot lesions during fixed orthodontic appliance treatment: A meta-analysis. J Int Soc Prev Community Dent. 2015 Nov-Dec;5(6):433-9. doi: 10.4103/2231-0762.167719. PMID 26759794
- [Background] Shimpo Y, Nomura Y, Sekiya T, Arai C, Okada A, Sogabe K, Hanada N, Tomonari H. Effects of the Dental Caries Preventive Procedure on the White Spot Lesions during Orthodontic Treatment-An Open Label Randomized Controlled Trial. J Clin Med. 2022 Feb 6;11(3):854. doi: 10.3390/jcm11030854. PMID 35160305
- [Background] Martignon S, Ekstrand KR, Lemos MI, Lozano MP, Higuera C. Plaque, caries level and oral hygiene habits in young patients receiving orthodontic treatment. Community Dent Health. 2010 Sep;27(3):133-8. PMID 21046903
- [Background] Chapman JA, Roberts WE, Eckert GJ, Kula KS, Gonzalez-Cabezas C. Risk factors for incidence and severity of white spot lesions during treatment with fixed orthodontic appliances. Am J Orthod Dentofacial Orthop. 2010 Aug;138(2):188-94. doi: 10.1016/j.ajodo.2008.10.019. PMID 20691360
- [Background] Ogaard B, Rolla G, Arends J. Orthodontic appliances and enamel demineralization. Part 1. Lesion development. Am J Orthod Dentofacial Orthop. 1988 Jul;94(1):68-73. doi: 10.1016/0889-5406(88)90453-2. PMID 3164585
- [Background] Tufekci E, Dixon JS, Gunsolley JC, Lindauer SJ. Prevalence of white spot lesions during orthodontic treatment with fixed appliances. Angle Orthod. 2011 Mar;81(2):206-10. doi: 10.2319/051710-262.1. PMID 21208070
- [Background] Fejerskov O. Concepts of dental caries and their consequences for understanding the disease. Community Dent Oral Epidemiol. 1997 Feb;25(1):5-12. doi: 10.1111/j.1600-0528.1997.tb00894.x. PMID 9088687
- [Background] Scheerman JFM, van Empelen P, van Loveren C, Pakpour AH, van Meijel B, Gholami M, Mierzaie Z, van den Braak MCT, Verrips GHW. An application of the Health Action Process Approach model to oral hygiene behaviour and dental plaque in adolescents with fixed orthodontic appliances. Int J Paediatr Dent. 2017 Nov;27(6):486-495. doi: 10.1111/ipd.12287. Epub 2017 Feb 7. PMID 28176383
- [Background] Scheerman JFM, van Meijel B, van Empelen P, Kramer GJC, Verrips GHW, Pakpour AH, Van den Braak MCT, van Loveren C. Study protocol of a randomized controlled trial to test the effect of a smartphone application on oral-health behavior and oral hygiene in adolescents with fixed orthodontic appliances. BMC Oral Health. 2018 Feb 7;18(1):19. doi: 10.1186/s12903-018-0475-9. PMID 29415697
- [Background] Rigau-Gay MM, Claver-Garrido E, Benet M, Lusilla-Palacios P, Ustrell-Torrent JM. Effectiveness of motivational interviewing to improve oral hygiene in orthodontic patients: A randomized controlled trial. J Health Psychol. 2020 Nov-Dec;25(13-14):2362-2373. doi: 10.1177/1359105318793719. Epub 2018 Sep 10. PMID 30198774
- [Background] Gao X, Lo EC, Kot SC, Chan KC. Motivational interviewing in improving oral health: a systematic review of randomized controlled trials. J Periodontol. 2014 Mar;85(3):426-37. doi: 10.1902/jop.2013.130205. Epub 2013 Jun 27. PMID 23805818
- [Background] Acharya S, Goyal A, Utreja AK, Mohanty U. Effect of three different motivational techniques on oral hygiene and gingival health of patients undergoing multibracketed orthodontics. Angle Orthod. 2011 Sep;81(5):884-8. doi: 10.2319/112210-680.1. Epub 2011 May 25. PMID 21612316
- [Background] Enaia M, Bock N, Ruf S. White-spot lesions during multibracket appliance treatment: A challenge for clinical excellence. Am J Orthod Dentofacial Orthop. 2011 Jul;140(1):e17-24. doi: 10.1016/j.ajodo.2010.12.016. PMID 21724067
- [Background] Ekstrand KR, Gimenez T, Ferreira FR, Mendes FM, Braga MM. The International Caries Detection and Assessment System - ICDAS: A Systematic Review. Caries Res. 2018;52(5):406-419. doi: 10.1159/000486429. Epub 2018 Mar 8. PMID 29518788
- [Background] Guarnizo-Herreno CC, Watt RG, Garzon-Orjuela N, Suarez-Zuniga E, Tsakos G. Health insurance and education: major contributors to oral health inequalities in Colombia. J Epidemiol Community Health. 2019 Aug;73(8):737-744. doi: 10.1136/jech-2018-212049. Epub 2019 May 16. PMID 31097482
- [Background] Marinho VC, Higgins JP, Sheiham A, Logan S. Fluoride toothpastes for preventing dental caries in children and adolescents. Cochrane Database Syst Rev. 2003;2003(1):CD002278. doi: 10.1002/14651858.CD002278. PMID 12535435
- [Background] Aljabaa A, McDonald F, Newton JT. A systematic review of randomized controlled trials of interventions to improve adherence among orthodontic patients aged 12 to 18. Angle Orthod. 2015 Mar;85(2):305-13. doi: 10.2319/031214-184.1. Epub 2014 Jul 21. PMID 25045779
- [Background] Gao X, Lo EC, McGrath C, Ho SM. Face-to-face individual counseling and online group motivational interviewing in improving oral health: study protocol for a randomized controlled trial. Trials. 2015 Sep 18;16:416. doi: 10.1186/s13063-015-0946-0. PMID 26385340
- [Background] Talic NF. Adverse effects of orthodontic treatment: A clinical perspective. Saudi Dent J. 2011 Apr;23(2):55-9. doi: 10.1016/j.sdentj.2011.01.003. Epub 2011 Jan 28. PMID 24151415